CLINICAL TRIAL: NCT04355039
Title: A Phase I Study of INCB053914 (Pan-PIM Kinase Inhibitor) and Pomalidomide With Dexamethasone in Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: INCB053914 and Pomalidomide With Dexamethasone for Relapsed and/or Refractory Multiple Myeloma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated for lack of funding.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Binod Dhakal, Assistant Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT-Dhakal-INCB053914
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Refractory Multiple Myeloma; Relapse Multiple Myeloma
Keywords: Multiple Myeloma; Refractory Multiple Myeloma; Relapse Multiple Myeloma; INCB053914; pan-PIM Kinase Inhibitor
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; Dexamethasone; Calcium Dobesilate; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pomalidomide, Dexamethasone & INCB053914 50 mg twice daily (Experimental): INCB053914 will have a dose escalation in a 3 + 3 design.
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: INCB053914 50 mg bis in die (BID)
- Pomalidomide, Dexamethasone & INCB053914 65 mg twice daily (Experimental): INCB053914 will have a dose escalation in a 3 + 3 design.
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: INCB053914 65 mg BID
- Pomalidomide, Dexamethasone & INCB053914 80 mg twice daily (Experimental): INCB053914 will have a dose escalation in a 3 + 3 design.
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: INCB053914 80 mg BID

INTERVENTIONS:
Drug: Pomalidomide — 4 mg Days 1-21
  Other Names: Pomalyst
Drug: Dexamethasone — 40 mg Days 1, 8, 15 and 22
  Other Names: Ozurdex
Drug: INCB053914 50 mg bis in die (BID) — Dose level 0: 50 mg BID
  Other Names: pan-PIM Kinase Inhibitor
  Arms: Pomalidomide, Dexamethasone & INCB053914 50 mg twice daily
Drug: INCB053914 65 mg BID — Dose level 1: 65 mg BID
  Other Names: pan-PIM Kinase Inhibitor
  Arms: Pomalidomide, Dexamethasone & INCB053914 65 mg twice daily
Drug: INCB053914 80 mg BID — Dose level 2: 80 mg BID
  Other Names: pan-PIM Kinase Inhibitor
  Arms: Pomalidomide, Dexamethasone & INCB053914 80 mg twice daily

SUMMARY:
This is a prospective, single-center, open-label phase Ib study aimed at determining a recommended phase II dose of INCB053914 and pomalidomide with dexamethasone. The trial will follow a 3 + 3 phase I dose-escalation design.

DETAILED DESCRIPTION:
This is a prospective, single-center phase I clinical study aimed at determining the maximum-tolerated dose and safety of INCB053914 (pan-PIM kinase inhibitor) and pomalidomide with dexamethasone in patients with relapsed and/or refractory multiple myeloma. Three candidate dose levels of INCB053914, 50 mg, 65 mg, and 80 mg twice daily will be considered.

The research team will utilize a 3+3 design to determine a safe dose of INCB053914 combined with fixed doses of pomalidomide (4 mg Days 1- Days 21) and dexamethasone (40 mg Days 1, 8, 15, 22).

The first three patients will be treated with INCB053914 twice daily at a dose of 50 mg.

Dose-limiting toxicity (DLT) assessment during the first 28-day cycle will be the basis for maximum-tolerated dose assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
2. Patient should have received ≥2 lines of therapy including at least two consecutive cycles of lenalidomide and a proteasome inhibitor alone or in combination and should be relapsed and/or refractory to lenalidomide and a proteasome inhibitor.
3. Measurable disease as defined (at least one of the following):

   * Serum M-protein level ≥0.5 g/dl or urine M-protein level ≥200 mg/24 hours. OR
   * Light chain multiple myeloma without measurable disease in the urine: serum Ig free light chain (FLC) ≥10 mg/dL and abnormal serum Ig kappa/lambda FLC ratio.
   * Non-secretory multiple myeloma (MM) with bidimensionally measurable plasmacytoma.
4. Male or female subjects ≥18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
6. Female subjects must meet one of the following:

   * Postmenopausal for at least one year before enrollment, OR
   * Surgically sterile (i.e., undergone a hysterectomy or bilateral oophorectomy), OR
   * If subject is of childbearing potential (defined as not satisfying either of the above two criteria), agrees to practice two acceptable methods of contraception (combination methods require use of two of the following: diaphragm with spermicide, cervical cap with spermicide, contraceptive sponge, male or female condom, hormonal contraceptive) from the time of signing of the informed consent form through 21days after the last dose of study agent, OR o Agrees to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable contraception methods.)
7. Male subjects, even if surgically sterilized (i.e., status postvasectomy), must agree to one of the following:

Practice effective barrier contraception during the entire study period and through 90 calendar days after the last dose of study agent, OR

o Agrees to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods] and withdrawal are not acceptable methods of contraception.)

Exclusion Criteria:

1. Prior use of PIM kinase inhibitors.
2. Prior pomalidomide refractory patients (last prior therapy was pomalidomide-containing regimen and/or patients within three months of pomalidomide dose).
3. Diagnosed or treated for malignancy other than multiple myeloma, except:

   * Malignancy treated with curative intent and with no known active disease present for ≥2 years before enrollment.
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   * Adequately treated carcinoma in situ (e.g., cervical, breast) with no evidence of disease.
4. Exhibiting clinical signs of meningeal or central nervous system involvement by multiple myeloma.
5. Known to be seropositive for human immunodeficiency virus, known to have hepatitis B surface antigen positivity, or known to have a history of hepatitis C.
6. Concurrent medical condition or disease (e.g., active systemic infection) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study. Specifically, any potential subject who is unsuitable for autologous stem cell transplant (ASCT) would be excluded from the study.
7. Clinically significant cardiac disease, including:

   * Myocardial infarction within six months before Cycle 1, Day 1, or unstable or uncontrolled disease/condition related to or affecting cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV).
   * Uncontrolled cardiac arrhythmia (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE] Version 5 grade 2 or higher) or clinically significant electrocardiogram (ECG) abnormalities.
   * Screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >470 msec.
8. Any of the following laboratory test results during the screening phase:

   * Absolute neutrophil count <1.0 × 109/L; no granulocyte-colony stimulating factor (G-CSF) treatment in the past seven days are allowed.
   * Hemoglobin level ≤7.5 g/dL (≤5 mmol/L); blood transfusions to maintain hemoglobin >7.5 g/dL are acceptable.
   * Platelet count <50 × 109/L for subjects in whom <50% of bone marrow nucleated cells are plasma cells; otherwise platelet count <50 × 109/L; no platelet transfusions in the past seven days are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
The number of subjects with dose-limiting toxicities. | 28 days
  The safety of INCB053914 with pomalidomide and dexamethasone in participants with relapsed and/or refractory multiple myeloma.

SECONDARY OUTCOMES:
The recommended phase II dose of INCB053914. | 28 days
  Based on number of dose-limiting toxicities.
Progression-free survival. | 2 Years
  This measure is the number of months participants remain free from evidence of disease. This will be captured using International Myeloma Working Group criteria.
Overall survival. | 2 Years
  Overall survival is defined from the number of months from initiation of treatment until death due to any cause. Participants without an observed progression / death event will be censored at the last follow-up or end of study.
Duration of response. | 2 Years
  The number of months from the date of first documented response (complete or partial) to the time of the next relapse/progression. This will be captured using International Myeloma Working Group criteria.
Efficacy of bone protective effect of INCB053914 in combination with pomalidomide and dexamethasone in patients with relapsed and/or refractory multiple myeloma. | 7 months
  The number of subjects with negative serum C terminal telopeptide type-X (CTX). This is determined by a blood draw.
The bone protective effect of INCB053914 in combination with pomalidomide and dexamethasone in patients with relapsed and/or refractory multiple myeloma. | 7 months
  The number of subjects with positive serum N terminal propeptide of procollagen (P1NP). This is determined by a blood draw.
The number of subjects with reduction of osteolytic lesions. | 7 months
  This will be determined by positron emission tomography (PET) /MRI scans, using RECIST.
The number of subjects with reduction of sclerosis formation. | 7 months
  This will be determined by positron emission tomography (PET) /MRI scans, using RECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Binod Dhakal, MD, Principal Investigator — Medical College of Wisconsin

IPD SHARING:
Plan to Share IPD: No